CLINICAL TRIAL: NCT04655365
Title: Detection and Monitoring of Metastasis by 18F-DCFPyL PET/CT in Subjects Starting Enzalutamide for Untreated Castration Resistant Prostate Cancer and Negative, Equivocal, or Oligometastatic Disease on Conventional Imaging (PROSTEP-002)
Brief Title: Detecting Metastases by PyL PET/CT in Subjects Starting Enzalutamide for Untreated Castration Resistant Prostate Cancer.
Acronym: PROSTEP-002
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROSTEP-002
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Untreated Castration Resistant Prostate Cancer; 18F-DCFPyL; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resistant Prostate Cancer and Negative, Equivocal or Oligometastatic Disease on Conventional Imaging (Experimental): Enrolled subjects will receive a single dose of 9 mCi (333 MBq) 18F-DCFPyL Injection followed by a single PET/CT scan acquired at 1-2 hours post-dosing. After initial 18F-DCFPyL PET/CT, the patients with positive 18F-DCFPyL PET/CT imaging will be treated with enzalutamide (160 mg po id) for M0CRPC disease within less than two weeks. 18F-DCFPyL PET/CT scan will then be repeated 90 days after the start of enzalutamide treatment.
  A final follow-up imaging (18F-DCFPyL PET/CT) at progression or at the final follow-up imaging examination at 18 months after the new complete ICF or in September 2026 (whichever comes first) will be performed.
  Interventions: Drug: Enzalutamide capsule

INTERVENTIONS:
Drug: Enzalutamide capsule — 160 mg po id
  Other Names: Xantdi

SUMMARY:
This study aimed to evaluate the diagnostic performance of 18F-DCFPyL (PyL) PET/CT in subjects presenting not previously treated for castration resistant prostate cancer and showing negative or equivocal findings per institutional standard of care conventional imaging

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common solid organ cancer in North American men and is initially androgen sensitive. Therefore, castration and/or androgen receptor blockade remains the central palliative treatment once PCa has metastasized or failed to locoregional therapies. Because androgen deprivation therapy is not curative, all patients will eventually progress to the metastatic castration-resistant prostate cancer state. About 5% of prostate cancers will be metastatic by conventional imaging techniques at diagnosis while most patients achieving CRPC state will first be localized and then progress to metastatic state later in the disease course. Therefore, a significant proportion of patients will progress through an intermediary state of disease defined as the non-metastatic CRPC state (M0CRPC). Over the last year and a half, M0CRPC treatment landscape has completely changed with demonstrating the benefits of second-generation antiandrogens (darolutamide, enzalutamide and apalutamide) to prevent progression of M0CRPC patients. Enzalutamide have then been approved by the Federal Drug Administration and Health Canada for the treatment of M0CRPC.

On the other hand, conventional imaging techniques based on bone turnover (bone scan (BS)) or anatomical features (magnetic resonance imaging (MRI) or computed tomography (CT)) have important limitations and poor accuracy. Bone scans (BS) is the commonest imaging technique used to detect bone metastases in the clinics. BS does not image directly cancer cells, but the effect of cancer on the bone. Other pathologies such as fractures, degenerative arthritis and other benign bone lesions can also cause focal uptake on BS and lead to false-positive results. Another drawback of BS is its poor sensitivity to image small metastases confined to bone marrow. These limitations stress the importance to improve PCa imaging by using new imaging modalities.

Because novel agents targeting the androgen synthesis and receptor axis (e.g. enzalutamide), bone metastasis (radium-223) and microtubules assembly (docetaxel, cabazitaxel) have been shown to increase metastatic CRPC patients overall survival, a burning question is to determine if the non-metastatic CRPC status is real. There is growing evidence that newer imaging techniques using positron emission tomography can improve metastasis detection accuracy and may refine PCa patient prognostic stratification and treatment eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate per original diagnosis, with undergoing androgen deprivation therapy such as prior bilateral orchiectomy or surgical castration or LHRH-agonists/LHRH-antagonists.
* Suspected recurrence of prostate cancer based on rising PSA under androgen deprivation therapy. Recurrent castration resistant prostate cancer patients are defined by a rising PSA >1 ng/mL under ADT or surgical castration and with testosterone castration levels < 1.7 nM (PCWG3 criteria).
* Negative, equivocal findings or oligometastatic disease (< 5) for prostate cancer on conventional imaging bone scan AND 2) abdomen-pelvis CT/MRI and chest CT or FDG-PET/CT or 18F-NaF PET/CT performed as standard of care workup within 90 days of signing the ICF.
* The subject is candidate for second line androgen axis targeted inhibitors such as enzalutamide and planned to receive it.
* Life expectancy ≥6 months as determined by the investigator
* Able and willing to provide signed informed consent and comply with protocol requirement
* PSA doubling time less or equal to 10 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
* Able to swallow the study drug and comply with study requirements.

Exclusion Criteria:

* Subjects administered any high energy (>300 KeV) gamma-emitting radioisotope within 5 physical half-lives prior to study drug injection.
* Receipt of investigational drug therapy for prostate cancer within 60 days of Day 1.
* Known or suspected brain metastasis or active leptomeningeal disease.
* Prior cytotoxic chemotherapy, aminoglutethimide, ketoconazole, abiraterone acetate, or enzalutamide for prostate cancer.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma). History of loss of consciousness (unless of cardiac origin) or transient ischemic attack within 12 months before enrollment.
* Major surgery within 4 weeks before randomization date.
* Absolute neutrophil count < 1000/μL, platelet count < 100,000/μL, or hemoglobin < 10 g/dL (6.2 mmol/L) at screening.
* Total bilirubin ≥ 1.5-times the upper limit of normal or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5-times the upper limit of normal at screening.
* Creatinine > 2 mg/dL (177 μmol/L) at screening.
* Albumin < 3.0 g/dL (30 g/L) at screening.
* Clinically significant cardiovascular disease
* Gastrointestinal disorder affecting absorption.
* Ongoing drug or alcohol abuse as per investigator judgment.
* Subject has received any investigational radioactive agent within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subjects with any medical condition or other circumstances that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completing the study.
* Contraindication to enzalutamide
* Treatment with specific (5-α reductase inhibitors, estrogens, cyproterone actetate, biologic agents with antitumor activity, systemic glucocorticoids, androgens, ...) within 4 weeks of day 1 and during the study treatment period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Determine the percentage of patients presenting new metastatic lesions detected by 18F-DCFPyL-PSMA PET/CT in castration resistant prostate cancer patients presenting non metastatic, equivocal or oligometastatic (< 5 metastasis) disease | Through study completion, an average of 1 year
  Number of patients presenting with metastases per compartment (bone, visceral, lymph node) determined by 18F-DCFPyL-PSMA PET/CT that were negative or equivocal on conventional imaging. determined by 18F-DCFPyL-PET/CT.
Determine the number of discordant lesions between conventional and PSMA-PET/CT imaging in castration resistant prostate cancer patients presenting with non metastatic, equivocal or oligometastatic (< 5 metastasis) disease defined by conventional imagi | through study completion, an average of 1 year
  Number of metastases per compartment (bone, visceral, lymph node) that are discordant between conventional imaging and 18F-DCFPyL-PSMA -PET/CT.
Determine the percentage of patients showing 18F-DCFPyL-PSMA PET/CT active lesions at progression (V5) that were active on either baseline and 3-month PSMA-PET/CT (extension phase) | through study extension phase completion, an average of 1 year
  At V5, number of patients presenting with metastases determined by 18F-DCFPyL-PSMA PET/CT that were active on either baseline and 3-month PSMA-PET/CT
In patients with 18F-DCFPyL-PSMA PET/CT active lesions at progression (V5), determine the percentage of lesions that were NOT active on either baseline and 3-month PSMA-PET/CT (New lesions) (extension phase) | through study extension phase completion, an average of 1 year
  Number of metastases per compartment (bone, visceral, lymph node) at V5 imaging that were NOT active on either baseline and 3-month PSMA-PET/CT.
  Number of metastases per compartment (bone, visceral, lymph node) that were active on either baseline and 3-month PSMA-PET/CT.

SECONDARY OUTCOMES:
Determine the intrapatient and interpatient 18F-DCFPyL-PSMA response rates defined by a 50% decrease in intralesional 18F-DCFPyL-PSMA uptake or 50% decrease in sum metastasis 18F-DCFPyL-PSMA uptake after 3 months of enzalutamide. | At the end of study completion, an average of 2 years
  Determine the changes in 18F-DCFPyL-PSMA sum metastasis SUVmax (or any other radiomic PET parameter) for each patient and the changes of 18F-DCFPyL-PSMA SUVmax (or any other radiomic PET parameter) in each lesion after 3 months of enzalutamide.
Determine the impact of 18F-DCFPyL-PSMA PET/CT at progression (V5) on patient's management. (Extension phase) | through study extension phase completion, an average of 1 year
  Management plan prior and after the last 18F-DCFPyL-PSMA PET/CT (V5)
In non-progressive patients defined by stable PSA, determine the percentage of patients showing active 18F-DCFPyL-PSMA PET/CT lesions at V5. (extension phases) | through study extension phase completion, an average of 1 year
  Number of patients presenting active 18F-DCFPyL-PSMA PET/CT lesions at V5 (among those who have not progressed).
Determine how 18F-DCFPyL-PSMA PET/CT radiomics at baseline or 3 months after enzalutamide start can predict time to biochemical progression under enzalutamide. (extension phase) | through study extension phase completion, an average of 1 year
  Metastases SUVmax (or any other radiomics PET parameter) for each patient at baseline (V1) and 3 months after enzalutamide start (V3). Date of enzalutamide start and of biochemical progression

OTHER OUTCOMES:
Number and sites of new lesions detected by 18F-DCFPyL-PSMA PET/CT at several PSA thresholds | At the end of study completion, an average of 2 years
  Number of metastasis per compartment (bone, visceral, lymph node) determined by 18F-DCFPyL-PET/CT when PSA is <1 ng/mL, 1 to 5 ng/mL and > 5 ng/mL.
Determine the percentage of patients showing metastatic lesions with enough 18F-DCFPyL uptake (above that of the liver) to justify radioligand therapy before and 3 months after enzalutamide treatment. | At the end of study completion, an average of 2 years
  Analyze if a patient shows one or several lesions with a 18F-DCFPyL uptake more than that of the liver.
Determine clinical and radiomics criteria to distinguish patients presenting with flares at 3-months (visit 3) from those that had real progression at V5. (Extension phase) | through study extension phase completion, an average of 1 year
  Clinical and radiomics characteristics of patients that had ≥1 progressive lesion on visit 3 DCFPyL-PSMA PET/CT but sustained PSA-response for up to six months which defines a flare phenomena (section 15.4.2)
Determine the percentage of patients with oligo-progressive (<5 sites) disease based on 18F-DCFPyL-PSMA PET/CT at V5 (extension phase) | through study extension phase completion, an average of 1 year
  Number of patients presenting with oligo-progressive (<5 sites) disease based on 18F-DCFPyL-PSMA PET/CT at V5.
Compare number of lesions determined by most recent conventional imaging (bone scintigraphy and CT-scan) with that of 18F-DCFPyL-PSMA PET/CT at V5 (extension phase) | through study extension phase completion, an average of 1 year
  Number of lesions per compartment (bone, visceral, lymph node) at V5 and the most recent conventional imaging and at 18F-DCFPyL-PSMA PET/CT at V5

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Pouliot, MD, Principal Investigator — CHU de Québec-Université Laval
Locations (4):
- Canada (4):
  - CHUM, Montreal, Quebec
  - CUSM, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No